CLINICAL TRIAL: NCT05212103
Title: PET Imaging of Cancer Patients Using 68Ga-DOTA-Siglec-9
Acronym: CANSI
Status: Enrolling by invitation | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1301/2022
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia; Melanoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum for determination of soluble VAP-1 level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a scientific study to determine expression of vascular adhesion protein 1 (VAP-1) in cancer patients by 68Ga-DOTA-Siglec-9 positron emission tomography/computed tomography (PET/CT) before and after cancer treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate expression of vascular adhesion protein 1 (VAP-1) in bone marrow and cancerous lesions before and after therapy using 68Ga-DOTA-Siglec-9 positron emission tomography/computed tomography (PET/CT). Patients with acute myeloid leukemia (AML) that undergo bone marrow transplantation and patients with melanoma and lung cancer that undergo chemotherapy will be studied. In addition, imaging results will be compared with clinical data and research data from blood samples. The study is of great clinical importance as other methods do not provide such comprehensive information on the presence of the VAP-1 molecule in the body, especially in the bone marrow and cancer tissue before and after cancer treatment. Research is also important for drug development targeting VAP-1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) and fit for allogeneic hematopoietic stem cell transplantation (alloHSCT), as assessed in the standard operating procedures.
* Diagnosis of metastatic melanoma and fit for immune checkpoint inhibitors or BRAF- and MEK inhibitors.
* Diagnosis of metastatic non-small cell lung cancer (NSCLC) (stage IV) and fit for immune checkpoint inhibitors and/or chemotherapy.
* Able and willing to give written informed consent and to comply with the study protocol.

Exclusion Criteria:

* Unsuitable for alloHSCT (AML), checkpoint inhibitors or BRAF- and MEK inhibitors (melanoma or checkpoint inhibitors and/or chemotherapy (NSCLC) according to the standard operating procedures.
* Unable or unwilling to comply with the study protocol for any reason.
* Evidence of significant uncontrolled concomitant diseases such as neurological, renal, hepatic, endocrine, or gastrointestinal disorders which, in the opinion of the Investigator, would preclude patient participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Turku University Hospital with acute myeloid leukemia (AML), metastatic melanoma and metastatic non-small cell lung cancer (NSCLC) (stage IV)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
68Ga-DOTA-Siglec-9 uptake in bone marrow and cancerous lesions | within a 1 day
  Standardized uptake value of PET tracer 68Ga-DOTA-Siglec-9 in the bone marrow and cancerous lesions

CONTACTS AND LOCATIONS:
Overall Officials: Anne Roivainen, Principal Investigator — Turku University Hospital, Turku PET Centre
Locations (1):
- Turku University Hospital, Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dadson P, Yla-Outinen H, Kalliokoski K, Tuokkola T, Malaspina S, Koivumaki M, Viitanen R, Rajala N, Silvoniemi M, Tolvanen T, Nuutila P, Jalkanen S, Saraste A, Saaresranta T, Taimen P, Roivainen A. Proof-of-concept PET imaging of pulmonary sarcoidosis using VAP-1-targeted radiotracer [68Ga]Ga-DOTA-Siglec-9. Respir Res. 2025 Dec 19. doi: 10.1186/s12931-025-03455-8. Online ahead of print. PMID 41420234